CLINICAL TRIAL: NCT06714591
Title: A Multicenter, Open-Label Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Preliminary Efficacy of BL-M11D1 in Patients With Relapsed/Refractory Acute Myeloid Leukemia.
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetic Profile, Efficacy of Bl-M11D1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-M11D1-HM-101
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label Phase 1 study to evaluate the safety, tolerability, pharmacokinetic profile, and initial efficacy of BL-M11D1 in subjects with relapsed/refractory acute myeloid leukemia (r/r AML). This study has two parts:
  Part 1: Dose Escalation Part 2: Dose Finding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Cohort A BL-M11D1 administered Days 1, 8 and 15 in 28-day cycle (Experimental): Cohort A: BL-M11D1 will be administered on Days 1, 8 and 15 by intravenous infusion every 28 days.
  Interventions: Drug: BL-M11D1
- Experimental: Cohort B BL-M11D1 administered Days 1, 4 7 or 8 in 28-day cycle (Experimental): Cohort B: BL-M11D1 will be administered on Days 1,4, 7 or 8 by intravenous infusion every 28 days.
  Interventions: Drug: BL-M11D1

INTERVENTIONS:
Drug: BL-M11D1 — The study includes 2 parts:
  Part 1 Dose escalation and Dose Finding

SUMMARY:
The objective of this study to evaluate the safety, tolerability, pharmacokinetic profile, and preliminary efficacy of BL-M11D1 in patients with relapsed/refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
BL-M11D1-HM-101 is a multi-center, Phase 1 study to evaluate the safety, tolerability, pharmacokinetic profile, and preliminary efficacy of BL-M11D1 in patients with relapsed/refractory acute myeloid leukemia.

This study will be conducted in two parts (dose escalation, and dose finding). Cohort A will be dosed on Days 1, 8,15 of a continuous 28-day treatment cycle. The cohort has different dose groups. Cohort B will be dosed on Days 1, 4, 7 or 8 of a continuous 28-day treatment cycle. The cohorts have different dose groups.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent
2. Age ≥18 years
3. Has a life expectancy of ≥3 months
4. Relapsed and/or refractory CD33-positive AML as determined by local pathology review that has failed initial standard of care therapy. Diagnosis of primary AML or AML secondary to myelodysplastic syndromes. Relapsed or refractory status. CD33-positive as confirmed by local flow cytometry or cytology
5. Has an Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 2
6. Toxicity of previous anticancer therapy has returned to Grade ≤1 as defined by NCI CTCAE V5.0, except for alopecia and endocrinopathies controlled by replacement therapy that must be Grade ≤2
7. Has adequate liver and renal function before registration, defined as: a. Hepatic function: Total bilirubin (TBIL) ≤1.5×ULN (≤3×ULN for subjects with Gilbert's syndrome), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN b. Renal function: Creatinine clearance ≥50 mL/min (Cockcroft-Gault, Chronic Kidney Disease Epidemiology Collaboration [CKD-Epi], or Modification of Diet in Renal Disease Study [MDRD] equations)
8. Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception during the course of the study and for 7 months after the last dose of study treatment. An additional contraceptive method, such as a barrier method (eg, condom), is recommended
9. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and must be nonlactating

Exclusion Criteria:

1. Subjects with acute promyelocytic leukemia (APL) or chronic myelogenous leukemia in blast crisis (CML)
2. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, major surgery, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other anticancer therapy within 2 weeks) prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration, or palliative radiotherapy within 2 weeks prior to the first administration
3. Subjects with history of severe heart disease, such as symptomatic congestive heart failure (CHF) ≥ Grade 2 (CTCAE 5.0), New York Heart Association (NYHA) ≥ Grade 2 heart failure, history of transmural myocardial infarction, unstable cardiac arrhythmias or angina pectoris within 6 months before screening
4. Subjects with prolonged QT interval (QTcF >470 msec), complete left bundle branch block, Grade 3 atrioventricular block or a history of additional risk factors for Torsades de Pointes (TdP; eg, heart failure as defined in Exclusion Criterion 3, chronic or recurrent hypokalemia that requires medical intervention, congenital long QT syndrome, family history of long QT syndrome) or any current concomitant medication known to prolong the QT/QTc interval or cause TdP
5. Active autoimmune diseases and inflammatory diseases, such as: systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc., except for Type I diabetes, hypothyroidism that can be controlled only by standard of care treatment, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis)
6. Subjects with other prior or concurrent malignancies except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after adequate resection, or other malignancy treated with curative intent with as disease-free interval of at least 1 year
7. Subjects with poorly controlled hypertension or uncontrolled hypertension by two or more antihypertensive drugs (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg)
8. Subjects with active acute or chronic graft vs. host disease (aGVHD or cGVHD) should be excluded from this study. Subjects with GVHD who are receiving treatment with systemic glucocorticoids >10 mg/day equivalent of prednisone should also be excluded from the study; however, treatment with low-dose glucocorticoids (≤10 mg/day equivalent of prednisone) is permitted
9. Subjects currently receiving immunosuppressive therapy should be excluded from this study.
10. Clinical evidence of disseminated intravascular coagulation (DIC). Smoldering low grade DIC is allowed after discussion with the sponsor
11. Subjects with stroke or transient ischemic attack (TIA) within 6 months before screening
12. Subjects with a thromboembolic event (eg, deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 6 months before screening except for those who are clinically stable and receiving treatment with adequate anticoagulant therapy for at least 3 weeks before screening
13. Subjects with active central nervous system (CNS) AML will be excluded. A lumbar puncture does not need to be performed unless there is clinical suspicion of CNS involvement per investigator judgment. Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS AML is allowed with the approval of the sponsor
14. Subjects with pre-existing ≥Grade 2 peripheral neuropathy
15. Subjects with advanced/ clinically significant lung diseases, such as poorly controlled COPD and asthma, restrictive lung disease, pulmonary hypertension etc.
16. Subjects who have a history of noninfectious interstitial lung disease (ILD)/ pneumonitis that required treatment with steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
17. Subjects who have a history of anaphylaxis or severe hypersensitivity to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of BL-M11D1
18. Subjects with known human immunodeficiency virus infection (HIV Ab positive) Subjects are allowed to participate if all of the following criteria are met: (1) Undetectable HIV RNA and CD4 count ≥350 cells/μL at screening, (2) No AIDS defining opportunistic infection within 12 months prior to screening, (3) On stable antiretroviral therapy (ART) for at least 4 weeks prior to screening with projected continuation of ART as clinically indicated while on the study
19. Subjects with active Hepatitis B virus (HBV) infection (positive HBsAg test). Subjects with chronic inactive HBV infection are eligible if they meet all of the following criteria:

    1. Have a HBV DNA viral load ≤ 500 IU/mL
    2. Have normal AST and ALT, OR if liver involvement is present, has AST and ALT <3 × ULN which are not attributed to HBV infection
    3. on antiviral treatment, as clinically indicated
20. Subjects with active Hepatitis C virus (HCV) infection (HCV antibody positive and HCV-RNA > the lower limit of detection). Subjects with a positive anti-HCV antibody are eligible only if PCR is negative for HCV RNA
21. Subjects with active or latent tuberculosis
22. Subjects with active and uncontrolled infections requiring IV antibiotic, antiviral, or antifungal treatment, such as severe pneumonia, bacteremia, sepsis, etc., within 1 week prior to first dose of study treatment. Subjects on stable oral antimicrobials with no clinical or laboratory evidence of active infection are eligible
23. Received an investigational drug within 2 weeks prior to first dose of study treatment.
24. Subjects who are pregnant, breastfeeding, or planning to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Participants with dose-limiting toxicities | 1 Year
  DLTs are defined as any of the following events that are not clearly due to the underlying disease, disease progression, or extraneous causes:
  * Any treatment-emergent adverse event (TEAE) of ≥ Grade 3 except those due to disease progression or extraneous cause
  * Any TEAE that leads to dose reduction or withdrawal Nonhematologic toxicities
  * Death
  * Hy's law cases
  * Grade ≥3 nonhematologic toxicities (with exceptions) Hematologic toxicity
  * Grade 4 thrombocytopenia or neutropenia lasting >42 days in the absence of persistent leukemia
  * Grade ≥3 platelet count decreased with clinically significant hemorrhage
Participants with Serious Adverse Events (SAEs) and treatment-emergent adverse events (TEAEs) | 1 Year
  Measuring the number of patients with serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs)
To determine the minimum safe and effective dose (MSED), maximum tolerated dose (MTD) if reached, and maximum administered dose (MAD) of BL-M11D1 in AML | 1 Year
  Determine the highest BL-M11D1 dose level at which ≤33% subjects experience a DLT during the DLT evaluation period and highest BL-M11D1 dose administered in the event and MTD cannot be defined.

SECONDARY OUTCOMES:
Cmax of BL-M11D1 | 1 Year
  Calculate maximum (peak) observed concentration of BL-M11D1
Tmax of BL-M11D1 | 1 Year
  Calculate time of maximum observed concentration of BL-M1D1
Tmax of free payload ED-04 | 1 Year
  Calculate time of maximum observed concentration of free payload ED-04
Cmax of free payload ED-04 | 1 Year
  Calculate maximum (peak) observed concentration of free payload ED-04
AUC(0-8) of BL-M11D1 | 1 Year
  Calculate area under the serum concentration-time curve of BL-M11D1 from time 0 to 8 hours
AUC(0-8) of free payload ED-04 | 1 Year
  Calculate area under the serum concentration-time curve of free payload ED-04 from time 0 to 8 hours
AUC(last) of BL-BM11D1 | 1 Year
  Calculate area under the serum concentration-time curve up of BL-M11D1 to the last quantifiable time
AUC(last) of free payload ED-04 | 1 Year
  Calculate area under the serum concentration-time curve up of free payload ED-04 to the last quantifiable time
Tmax of anti-CD33 antibody | 1 Year
  Calculate time of maximum observed concentration of anti-CD33 antibody
AUC (0-8) of anti-CD33 antibodies | 1 Year
  Calculate area under the serum concentration-time curve of anti-CD33 antibodies from time 0 to 8 hours
AUC (last) anti-CD33 antibodies | 1 Year
  Calculate area under the serum concentration-time curve up of anti-CD33 antibodies to the last quantifiable time
Overall Response Rate (ORR) | 1 Year
  To assess the clinical efficacy of BL-M11D1 as measured by ORR using RECIST criteria v 1.1
Duration of response (DOR) | 1 Year
  To access the clinical efficacy of BL-M11D1 as measured by DOR using RECIST criteria 1.1
Complete Remission (CR) | 1 Year
  To assess the anti-cancer activity of BL-M11D1 as measured by CR using the European LeukemiaNet (ELN) 2022 AML criteria.
CR with partial hematologic recovery (CRh) | 1 Year
  To assess the anti-cancer activity of BL-M11D1 as measured by CR using the European LeukemiaNet (ELN) 2022 AML criteria.
CR with incomplete hematologic recovery (CRi) | 1 Year
  To assess the anti-cancer activity of BL-M11D1 as measured by CR using the European LeukemiaNet (ELN) 2022 AML criteria.
CR/CRi, CRs with or without measurable residual disease (MRD) | 1 Year
  To assess the anti-cancer activity of BL-M11D1 as measured by CR using the European LeukemiaNet (ELN) 2022 AML criteria.
morphologic leukemia-free state (MLFS) | 1 Year
  To assess the anti-cancer activity of BL-M11D1 as measured by CR using the European LeukemiaNet (ELN) 2022 AML criteria.
partial remission (PR) | 1 Year
  To assess the anti-cancer activity of BL-M11D1 as measured by CR using the European LeukemiaNet (ELN) 2022 AML criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Loren VanPelt, Study Director — SystImmune Inc.
Locations (14):
- United States (14):
  - City of Hope, Duarte, California
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - Yale Cancer Center, Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - START Midwest/The Cancer and Hematology Center, Grand Rapids, Michigan
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - WVCI Oncology Associates of Oregon, Eugene, Oregon
  - SCRI -TriStar BMT, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology, P.A., San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No